CLINICAL TRIAL: NCT02019017
Title: Endoscopic Block of the Sphenopalatine Ganglion With Botulinum Toxin in Intractable Cluster Headache - Safety Issues
Brief Title: Botox Injection in Treatment of Cluster Headache
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTACH2012; 2012-000248-91 (EudraCT Number)
Record Dates: First submitted 2013-11-21; First posted 2013-12-24 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Cluster Headache
Keywords: Cluster Headache; Botulinum Toxin Type A; Sphenopalatine Ganglion Block; Autonomic Nerve Block
MeSH Terms: conditions — Cluster Headache | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum Toxin Type A 25 IU (Experimental): The first five patients will be injected 25 IU of Botulinum Toxin Type A
  Interventions: Drug: Botulinum Toxin Type A 25 IU
- Botulinum Toxin Type A 50 IU (Experimental): the next five patients will receive 50 IU of Botulinum Toxin Type A
  Interventions: Drug: Botulinum Toxin Type A 50 IU

INTERVENTIONS:
Drug: Botulinum Toxin Type A 25 IU
  Other Names: Botox
  Arms: Botulinum Toxin Type A 25 IU
Drug: Botulinum Toxin Type A 50 IU
  Other Names: Botox
  Arms: Botulinum Toxin Type A 50 IU

SUMMARY:
Cluster headache is an intense and powerful, one-sided headache accompanied by involuntary symptoms such as red eye, droopy eyelids, flow of tears, small pupils and one-sided facial sweating. The headache is believed to be the most intense of all headaches and among many is totally disabling and of great personal and social consequences. For a small group of patients with episodic and most chronic form, drug therapy has little effect. For them, surgery can be a solution.

Neuroradiology has found evidence of a possible original activation of cluster headache from the portion of the brain called hypothalamus. Furthermore, an activation of the parasympathetic nervous system through the sphenopalatine ganglion, which may also explain some of the one-sided involuntary symptoms, is suspected in cluster headache. Injection of Botulinum toxin type A (BTA) inhibits secretion of synaptic acetylcholine resulting in nerve signals being blocked. The duration of such a blockade is believed to be 3-9 months.

The purpose of the present study is to develop and evaluate a new surgical procedure with injection of BTA for blocking of the sphenopalatine ganglion. The goal is to relieve the symptoms of refractory cluster headache with a minimal invasive procedure.

The main objective of the project is to determine the safety of BTA injection in the area of the sphenopalatine ganglion of refractory cluster headache and detect the adverse events. Secondary objectives are to identify the changes of headache attacks by the method used.

ELIGIBILITY:
Inclusion Criteria:

* Informed and written consent
* Cluster headaches defined in ICHD-2 criteria, duration of periods of attacks normally more than 2 months and insufficient effect of available prophylactic treatment

Exclusion Criteria:

* Heart or lung disease
* Any kind of systematic or local disease or illness that may significantly increase the risk of complications for the procedure, related to injection or anesthesia
* Psychiatric illness that hinders participation in the study
* Known pregnancy or breast feeding
* Inadequate use of contraceptives
* Overuse or abuse of opioids
* Abuse of medications, narcotics or alcohol
* Allergy or any other hypersensitivity reactions against marcain, lidocaine, xylocain or adrenalin, botulinum toxin type A, Botox or any of it's constituents or any other related medication
* Treatment with medication that can interact with botulinum toxin type A

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Safety aspects / Number of adverse events and number of participants with adverse events as a measure of safety | For the follow-up period of 6 months
  Number of adverse events and number of participants with adverse events after BTA injection in the area of the sphenopalatine ganglion and severity of adverse events. Registration of any adverse events categorized by probable relationship to drug, the surgical procedure or anesthesia. Data obtained from the headache diaries as well as open questions during consultations.

SECONDARY OUTCOMES:
Cluster headache attack frequency | Average number of attacks of baseline compared to average of week 3 and 4 after injection
Hours with cluster headache | Average of baseline compared to average of week 3 and 4 after injection
Days with cluster headache | Average of baseline compared to average of week 3 and 4 after injection

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F Bratbak, MD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Department of Neuroscience, Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Bratbak DF, Nordgard S, Stovner LJ, Linde M, Folvik M, Bugten V, Tronvik E. Pilot study of sphenopalatine injection of onabotulinumtoxinA for the treatment of intractable chronic cluster headache. Cephalalgia. 2016 May;36(6):503-9. doi: 10.1177/0333102415597891. Epub 2015 Jul 31. PMID 26232105